CLINICAL TRIAL: NCT01053221
Title: Mycophenolic Acid Monotherapy in Recipients of HLA-identical Living-Related Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding loss
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2005-0357; 2012-0343 (Other: HS-IRB)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Kidney Transplantation
Keywords: mycophenolate; living donor
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MPA monotherapy (Experimental): Subjects will discontinue calcineurin inhibitor (cyclosporine or tacrolimus) and remain on MPA (mycophenolate mofetil or mycophenolate sodium) monotherapy
  Interventions: Drug: Mycophenolic Acid
- Control: MPA and CNI (Active Comparator): Subjects will continue with their current immunosuppressive regimen of MPA (mycophenolate mofetil or mycophenolate sodium) and calcineurin inhibitor (cyclosporine or tacrolimus)
  Interventions: Drug: Standard of Care: CNI and MPA

INTERVENTIONS:
Drug: Mycophenolic Acid — Mycophenolate mofetil: 750mg po bid x 36 months OR mycophenolate sodium 540mg po bid x 36 months
  Other Names: cellcept, myfortic
  Arms: MPA monotherapy
Drug: Standard of Care: CNI and MPA — Tacrolimus or cyclosporine: dosed according to trough levels per standard of care Mycophenolate mofetil 750mg po bid or mycophenolate sodium 540mg po bid x 36 months
  Arms: Control: MPA and CNI

SUMMARY:
This randomized trial will enroll adult recipients of HLA-identical living kidney transplants who are at least 1 year post-transplant. All subjects will be taking Prograf (tacrolimus) or cyclosporine and mycophenolic acid (CellCept or Myfortic) and then be randomized (1:2) to either continue calcineurin inhibitors or to taper off of calcineurin inhibitors. The hypothesis is that mycophenolic acid monotherapy permits long-term rejection-free renal allograft function in the absence of long-term calcineurin inhibitors in this fully matched renal transplant cohort.

DETAILED DESCRIPTION:
The objective of the study is to safely move HLA-identical renal transplant recipients from 2 immunosuppressive drugs (calcineurin inhibitor and mycophenolic acid) to mycophenolic acid monotherapy. Safety will be assessed by monitoring renal function in subjects in the withdrawal group compared to those who remain on the standard 2-drug immunosuppression protocol. Results of immunological monitors such as DTH regulation in response to donor minor antigens and development of anti-donor antibodies will be correlated with successful withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-75 years of age.
* Subjects who are recipients of HLA-identical living donor renal allografts from a sibling and are at least 1 year post transplant, their donors and mothers.
* Subjects must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* GFR <40ml/min;
* diagnosis of SLE,
* Subjects with proteinuria (defined as a protein:creatinine ratio of >1 or an amount less than this deemed significant on an individual subject basis by the principal investigator),,
* multi-organ transplant;
* known hypersensitivity to, Prograf, Neoral, CellCept or Myfortic;
* history of documented post transplant non-compliance with medications, transplant clinic or laboratory follow-up;
* therapy with an investigational immunosuppressive drug within 6 weeks of study entry;
* history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study;
* patients on less than 500 mg PO BID of CellCept or 360 mg PO BID of Myfortic at the time of potential randomization,
* history of humoral rejection post transplant,
* maintenance or for cause treatment with steroids (prednisone) within 3 months of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Burlingham, PhD, Principal Investigator — University of Wisconsin, Madison; Hans Sollinger, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 16 enrolled participants,1 participant never got randomized and 1 participant did not show up for any of the appointments. Only 14 started in the study.
Period: Overall Study
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Started | 5 | 9
Completed | 0 | 0
Not Completed | 5 | 9
Not completed — The study was closed prematurely | 5 | 9

BASELINE CHARACTERISTICS:
Population: The study was closed prematurely and there is no data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | MPA Monotherapy | Control: MPA and CNI | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Kidney Allograft Rejection and Graft Loss
Time Frame: 36 months
Population: The study was closed prematurely. Data were not collected
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Renal Function Measured by Serum Creatinine and eGFR
Time Frame: 36 months
Population: The study was closed prematurely. No data was collected
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Incidences of Infection and Malignancy
Description: Number of incidences of infection and malignancy will be reported.
Time Frame: 36 months
Population: The study was closed prematurely. No data was collected
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient Survival
Description: patient survival
Time Frame: 36 months
Population: The study was closed prematurely. Data were not collected
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Trans-vivo Delayed Type Hypersensitivity (DTH) Assay
Description: Delayed type hypersensitivity (DTH) reactivity status to donor and minor antigens will be detected using trans-vivo DTH assay. This information will help determine if T-regulatory cells are present, and whether such cells predict outcome of Calcineurin inhibitor withdrawal.
Time Frame: 36 months
Population: The study was closed prematurely. Data were not collected
Arm/Group | MPA Monotherapy | Control: MPA and CNI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not monitored.
Arm/Group | MPA Monotherapy | Control: MPA and CNI
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No